CLINICAL TRIAL: NCT05103150
Title: Optical Enhancement Virtual Chromoendoscopy With High-definition Optical Magnification for Duodenal Mucosa Characterization in Coeliac Disease Patients.
Brief Title: Virtual Chromoendoscopy With Magnification in Coeliac Disease.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: IECED-10142021
Record Dates: First submitted 2021-10-15; First posted 2021-11-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Endoscopy; Gastrointestinal
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: High-definition white light endoscopy (HD-WLE) — Evaluation of the duodenal mucosa with HD-WLE (EG-29i10 gastroscope and EPKi7010 video processor). The endoscopy images will be seen on a 27inch, flat panel, high-definition LCD monitor (Radiance™ ultraSC-WU27-G1520 model) by one endoscopist, randomly assigned via esophagogastroduodenoscopy.
  There were used the following standard endoscopic findings were: a) "scalloping" or dented aspect of the duodenal folds; b) submucosal vascular pattern; c) "mosaicism" or micronodular look of the mucosa; d) grooves and fissurations of the mucosa.
Diagnostic Test: HD-WLE plus I-Scan optical enhancement (OE) virtual chromoendoscopy with High-definition optical magnification (HD-OM) — Evaluation of the duodenal mucosa through upper endoscopy with the OE System (EPK-i7010 HD Video Processor and MagniView™ EG-2990Zi Video Gastroscope) with intravenous sedation in a standardized manner. This technique involves using a distal black rubber hood (OE-A58; Pentax) at the tip of the endoscope, to fix the distance between the tip of the endoscope and the gastric mucosa at 2 mm. The OE System will be used in mode one and mode two without HD-OM to obtain an overview of the duodenal surface and identify any changes in the mucosa, then HD-OM will be implemented.
  There were used OE criteria as previously validated by Cammarota et al: brightness, Ave/peak, blue, red, surface, contrast, and tone enhancement.

SUMMARY:
High-definition white light endoscopy (HD-WLE) does not usually allow the visualization of duodenal villous patterns and may be inaccurate for assessing coeliac disease (CD). To the best of the knowledge of the authorship, there is no prospective study that has evaluated the accuracy of combining high-definition optical magnification (HD-OM) with i-Scan optical enhancement (OE) virtual chromoendoscopy for evaluation of duodenal villous patterns in the context of CD suspicion. Combining both techniques can also guide better duodenal biopsies. This study pursues to compare diagnostic accuracy between HD-WLE and HD-OM with OE using histology as the gold standard in detecting villous abnormalities in CD.

DETAILED DESCRIPTION:
High-definition white light endoscopy (HD-WLE) does not usually allow the visualization of duodenal villous patterns and may be inaccurate for assessing coeliac disease (CD). In addition, HD-WLE findings depend on CD severity. The lesser the disease severity, the higher possibility of showing a normal HD-WLE appearance. Thus, sampling routine duodenal biopsies have been suggested. However, this is time-consuming, expensive, and maybe excessive in low-risk groups. Sampling routine duodenal biopsies could also be unsuccessful, obtaining normal biopsies.

Novel endoscopic techniques have played an exciting role in increasing the accuracy of macroscopic evaluation of duodenal villous patterns. There have been described retrospective and prospective studies using chromoendoscopy, narrow-band imaging, optical coherence tomography, water immersion, confocal laser endomicroscopy, high-resolution magnification endoscopy, capsule endoscopy, and I-scan technology. However, results are disjunct, with no consensus.

The iSCAN optical enhancementTM (OE) System (PENTAX Medical, Tokyo, Japan) virtual chromoendoscopy has been developed to improve the blood vessels' visibility, ducts of the glands, and surface structures in addition to the traditional iSCAN functions. High-definition optical magnification (HD-OM) endoscopes have been developed and can combine HD imaging with OM to produce detailed images with a magnification of up to 136X. This imaging technique facilitates the evaluation of the superficial vascular aspects of the mucosa, enabling the identification of early signs of inflammation or lesions not previously seen with conventional endoscopy.

Prospective data have demonstrated that magnification endoscopy has superior diagnostic sensitivity in detecting villous atrophy compared to HD-WLE, being efficiently handled by all endoscopists. On another side, virtual chromoendoscopy has shown disjunct results across the literature. To the best of the knowledge of the authorship, there is no prospective study that has assessed the accuracy of combining HD-OM with i-Scan OE for evaluation of duodenal villous patterns in the context of CD suspicion. Combining both techniques can also guide better duodenal biopsies.

This study pursues to better characterize duodenal mucosa through OE with HD-OM in gluten-free diet (GFD) naïve patients with CD suspicion to correlate these findings with histology. As a second aim, to compare diagnostic accuracy between HD-WLE and HD-OM with OE using histology as the gold standard in detecting villous abnormalities in CD.

ELIGIBILITY:
Inclusion Criteria:

* Patients naïve to GFD;
* With clinical history suggestive of malabsorption (weight loss, chronic diarrhea, iron-deficiency, anemia, etc.);
* And serologic suspicion of CD as positive or borderline antiendomysial (normal values are absent for both IgA and IgG) and antitransglutaminase antibodies (normal values 0-10 U/mL).

Exclusion Criteria:

* Presence of severe gastrointestinal or systemic disease (e.g., chronic pancreatitis, liver cirrhosis, and blood coagulation disorders) impacts cardiovascular risk assessment.
* Presence of duodenal ulcer in the context of patients with upper gastrointestinal bleeding.
* History of any type of duodenal surgery.
* Pregnancy or nursing female.
* Refusal to participate in this observational trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, naïve to GFD, with clinical suspicion of CD who underwent endoscopic assessment.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Marsh's classification as revised by Oberhuber et al. | Six months
  Histology findings will be recorded and graded according to Marsh's classification as revised by Oberhuber et al (Marsh 0, Marsh 1, Marsh 2, Marsh 3a, Marsh 3b, and Marsh 3c). HD-WLE and HD-OM findings will be correlated with Marsh's classification. Finally, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) of HD-WLE and HD-OM will be calculated, considering Marsh's classification as gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, MD FASGE, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Raju SA, White WL, Lau MS, Mooney PD, Rees MA, Burden M, Ciacci C, Sanders DS. A comparison study between Magniview and high definition white light endoscopy in detecting villous atrophy and coeliac disease: A single centre pilot study. Dig Liver Dis. 2018 Sep;50(9):920-924. doi: 10.1016/j.dld.2018.03.037. Epub 2018 Apr 11. PMID 29807874
- [Result] Gadermayr M, Wimmer G, Kogler H, Vecsei A, Merhof D, Uhl A. Automated classification of celiac disease during upper endoscopy: Status quo and quo vadis. Comput Biol Med. 2018 Nov 1;102:221-226. doi: 10.1016/j.compbiomed.2018.04.020. Epub 2018 Apr 27. PMID 29739614
- [Result] Bonatto MW, Kotze L, Orlandoski M, Tsuchyia R, de Carvalho CA, Lima D, Kurachi G, Orso IR, Kotze L. Endoscopic evaluation of celiac disease severity and its correlation with histopathological aspects of the duodenal mucosa. Endosc Int Open. 2016 Jul;4(7):E767-77. doi: 10.1055/s-0042-108190. Epub 2016 Jun 29. PMID 27556094
- [Result] Iacucci M, Poon T, Gui XS, Subrata G. High definition i-SCAN endoscopy with water immersion technique accurately reflects histological severity of celiac disease. Endosc Int Open. 2016 May;4(5):E540-6. doi: 10.1055/s-0042-105955. Epub 2016 May 10. PMID 27227112
- [Result] Penny HA, Mooney PD, Burden M, Patel N, Johnston AJ, Wong SH, Teare J, Sanders DS. High definition endoscopy with or without I-Scan increases the detection of celiac disease during routine endoscopy. Dig Liver Dis. 2016 Jun;48(6):644-9. doi: 10.1016/j.dld.2016.02.009. Epub 2016 Feb 26. PMID 26995214
- [Result] Ianiro G, Gasbarrini A, Cammarota G. Endoscopic tools for the diagnosis and evaluation of celiac disease. World J Gastroenterol. 2013 Dec 14;19(46):8562-70. doi: 10.3748/wjg.v19.i46.8562. PMID 24379573
- [Result] De Luca L, Ricciardiello L, Rocchi MB, Fabi MT, Bianchi ML, de Leone A, Fiori S, Baroncini D. Narrow band imaging with magnification endoscopy for celiac disease: results from a prospective, single-center study. Diagn Ther Endosc. 2013;2013:580526. doi: 10.1155/2013/580526. Epub 2013 Aug 6. PMID 23983448